CLINICAL TRIAL: NCT07318649
Title: Phase 2 Clinical Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of GH21 Capsules Combined With D-1553 Tablets in Subjects With Locally Advanced or Metastatic Solid Tumors With the KRASG12C Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Genhouse Bio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GH21C204
Record Dates: First submitted 2025-12-19; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Masking Description: open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects received treatment with GH21 combined with D-1553, with 21 days as one cycle (Experimental): D-1553 tablet, BID, orally. Each cycle lasts 3 weeks. GH21 Capsule: QD, oral, Each treatment cycle lasts 3 weeks.
  Interventions: Drug: GH21，D-1553

INTERVENTIONS:
Drug: GH21，D-1553 — * D-1553 tablet, BID, orally. Each cycle lasts 3 weeks.
  * GH21 Capsule: QD, oral, Each treatment cycle lasts 3 weeks.

SUMMARY:
The study is divided into 2 cohorts, Cohort 1 is patients with KRASG12C mutated non-small cell lung cancer who have failed standard therapy or no standard therapy and have been treated with KRASG12C inhibitor; Cohort 2 is patients with KRASG12C mutated solid tumors (except non-small cell lung cancer) who have failed standard therapy or have no standard therapy and have been treated with KRASG12C inhibitor. Each cohort consists of two stages, and 10 subjects are planned to be enrolled in the first stage of each cohort. According to the preliminary efficacy and safety data, each party will discuss and decide whether to continue the second stage. Twenty to fifty subjects were planned to be enrolled in Stage II of each cohort. A total of 20-120 subjects were enrolled.

Screened eligible subjects received GH21 in combination with D-1553 in 21-day cycles until the investigator considered the subject no longer benefiting, or the subject developed intolerable toxicity, or the subject withdrew consent, or the subject died, or was lost to follow-up, or received a new anticancer treatment, whichever came first.

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients or their legal representatives can understand and voluntarily sign a written informed consent form (before starting this study and any study procedures); 2)Age ≥ 18 years, male or female; 3)Cohort 1: Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer with KRASG12C mutation who have failed standard therapy or no standard therapy and have been treated with KRASG12C inhibitors; Cohort 2: Histologically or cytologically confirmed locally advanced or metastatic solid tumors (except non-small cell lung cancer) with KRASG12C mutation who have failed standard therapy or have no standard therapy and have been treated with KRASG12C inhibitors.

  4)Patients must have at least one measurable lesion that meets the definition of RECISTv1.1 (tumor lesions located in previously irradiated areas or other locoregional treatment sites are generally not considered measurable unless there is definite progression of the lesion); 5)Expected survival ≥ 3 months; 6)ECOG performance score: 0-1; 7)Patients must have adequate organ function, defined as follows: Blood
  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L without granulocyte colony-stimulating factor support within 14 days;
  * Platelets≥100×109/L without thrombopoietin (TPO) and interleukin-11 (IL-11) transfusion within 14 days;
  * Hemoglobin ≥ 90 g/L without transfusion within 14 days and without erythropoietin (EPO); Renal
  * Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 60 ml/min calculated using the modified Cockcroft-Gault equation or eGFR ≥ 60 ml/min estimated by the MDRD equation; Liver
  * Albumin ≥ 3.0 g/dL;
  * Total bilirubin ≤ 1.5 × ULN; in case of liver metastasis, total bilirubin ≤ 2.5 × ULN;
  * AST/ALT ≤ 2.5 × ULN; in case of liver metastasis, AST/ALT ≤ 5 × ULN; Coagulation
  * International normalized ratio (INR) and prothrombin time (PT) ≤ 1.5 × ULN unless the patient is receiving anticoagulant therapy (INR < 2.5 × ULN) and PT or PTT is within the therapeutic range of the intended use of anticoagulants;
  * Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN unless the patient is receiving anticoagulant therapy (APTT < 2.5 × ULN) and PT or PTT is within the therapeutic range of the intended use of anticoagulants.

    8)Men of childbearing potential and women of childbearing potential must agree to practice reliable contraception (hormonal or barrier methods or abstinence) from signing of informed consent until 6 months after the last dose of study drug. Females of childbearing potential must have a negative pregnancy test ≤ 7 days prior to the first dose of study drug.

Exclusion Criteria:

* 1)Patients who have received chemotherapy, biological agents for anti-tumor therapy within 3 weeks before the first dose, radiotherapy, endocrine therapy and other anti-tumor drugs within 4 weeks before the first dose, except for the following:

  * nitrosourea or mitomycin C within 6 weeks before the first use of study drugs;
  * oral fluorouracil, small molecule targeted drugs and Chinese herbal medicine or Chinese patent medicine with anti-tumor indications within 5 half-lives or 2 weeks before the first use of study drugs (whichever is shorter);
  * Local palliative radiotherapy within 2 weeks before the first use of study drugs; 2)Receiving other unmarketed investigational drugs or treatments within 5 half-lives or 4 weeks (whichever is shorter) before the first dose; 3)Patients who underwent major organ surgery (excluding needle biopsy) or had significant trauma within 4 weeks before the first dose, or required elective surgery during the trial; 4)Use of strong inhibitors or strong inducers of CYP3A4 or P-gp within 2 weeks or 5 half-lives before the first dose; 5)Previous treatment with other SHP2 inhibitors. 6)Evidence of the following cardiac diseases: acute myocardial infarction, unstable angina pectoris, coronary artery bypass grafting, cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose;
  * Grade III-IV heart failure according to New York Heart Association functional classification at screening;
  * left ventricular ejection fraction (LVEF)≤50% by echocardiography (ECHO) at screening;
  * Fridericia-corrected QT interval (QTcF)≥450 ms (male) and≥470 ms (female) at screening;
  * poorly controlled hypertension (systolic blood pressure≥160 mmHg and/or diastolic blood pressure≥100 mmHg) after drug therapy at screening; 7)Dysphagia or gastrointestinal diseases or other malabsorption conditions affecting drug absorption, such as intestinal obstruction, Crohn 's disease, ulcerative colitis, short bowel syndrome, gastric emptying disorder or severe gastrointestinal related toxicity before the first dose and not recovered to less than grade 2; or confirmed to have clinically significant or acute gastrointestinal diseases; 8)Uncontrolled pleural effusion, pericardial effusion or pleural effusion requiring repeated drainage (once a month or more frequently); 9)Patients with active brain metastases or with symptoms of active central nervous system metastases including headache, vomiting and vertigo are eligible only if all of the following criteria are met, and asymptomatic patients with CNS lesions treated or untreated are eligible: • Measurable lesions located outside the CNS as determined by RECISTv1.1;
  * Stable brain metastases after treatment are defined as no evidence of disease progression or bleeding within 28 days before the start of treatment, and steroid hormones and other therapeutic agents are discontinued for at least 14 days before enrollment; 10)patients with interstitial pneumonia within 6 months before the first dose, or any evidence of clinically active interstitial lung disease; 11)Hyperarterial/venous thrombotic events within 6 months before the first dose, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis and pulmonary embolism; 12)Patients with a history of other malignant tumors (cured skin squamous cell carcinoma in situ, basal cell carcinoma and cervical carcinoma in situ that have not recurred for 5 years, unless the investigator believes that they can be enrolled; in the dose escalation stage, unless the investigator believes that they can be enrolled); 13)Patients who have a history of severe allergy, or have a history of allergy to test drugs/any excipients/combination therapy drugs, or have a history of allergy to multiple drugs; 14)Hepatitis B virus infection (HBsAg positive and DNA copy number > 1000 IU/ml); or hepatitis C virus infection (HCV antibody positive, HCV RNA > upper limit of normal); or human immunodeficiency virus infection (HIV antibody positive); 15)Active infection (≥ Grade 2) requiring anti-infective treatment or fever of unknown origin exceeding 38℃ within 28 days before the first dose; 16)autoimmune diseases in the active stage as judged by the investigator within 28 days prior to the first dose; 17)Any toxicity caused by previous anti-tumor treatment before the first dose has not recovered CTCAE 5.0 grade evaluation ≤ 1 (unless alopecia, grade 2 peripheral neuropathy and/or other adverse events ≤ grade 2 that do not pose a safety risk); 18)Pregnant or lactating women; 19)The investigator considers that there are any clinical or laboratory abnormalities or other reasons that make the subject unsuitable to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on RECIST 1.1 criteria | 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)

SECONDARY OUTCOMES:
Safety and tolerability | 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs , etc
Duration of response (DOR) based on RECIST 1.1 criteria | 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) based on RECIST 1.1 criteria | 2 years
  DCR is defined as proportion of participants with complete response, partial response, stable disease(CR+PR+SD).
Progression-free survival (PFS) based on RECIST 1.1 criteria | 2 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression or death which occurs first.
Overall survival (OS) | 2 years
  OS is defined as the interval of time between the date of first treatment until death, loss to follow up or termination of the study by the sponsor
Plasma concentration (Cmax) | 2 years
  Peak Plasma concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No